CLINICAL TRIAL: NCT00465634
Title: Screening for Placental Insufficiency by a Combination of Second Trimester Uterine Artery Doppler and Maternal Serum Leptin and Lipids
Brief Title: Doppler and Biological Second Trimester Placental Insufficiency Screening
Acronym: ARTULEP
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Pr Franck Perrotin, CHRU de Tours
Other Study IDs: PHRR02-FP/ARTULEP
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Pre-Eclampsia; Fetal Growth Retardation; Placental Insufficiency
Keywords: Screening; uterine artery Doppler; HELLP syndrome; abruption
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation; Placental Insufficiency; HELLP Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess the role of uterine artery and maternal serum leptin and lipids and their combination in screening for pre-eclampsia and small-for-gestational-age (SGA) fetuses at 20-24 weeks of gestation

DETAILED DESCRIPTION:
Pre-eclampsia (PE) and intrauterine growth restriction (IUGR) are known as major factors in perinatal morbidity and mortality. Routine antenatal care is focused on the detection of women at increased risk to apply this population a program of careful monitoring and appropriate intervention.

Uterine artery Doppler during anomaly scan at 20 to 24 weeks in selected women at increased risk, has proved to be accurate to detect those who will develop PE or IUGR during the second half of pregnancy. Studies have reported detection rate of 50-70% for a 5% false positive rate in women developing early pre-eclampsia.

A variety of proteins and hormones have been studied as potential markers for pre-eclampsia. Among these protein serum placental leptin has demonstrated higher levels in pregnant women who will subsequently develop pre-eclampsia. However, screening performance of leptin detection in early pregnancy has never been assessed.

Our study is aimed to evaluate the performance of serum leptin measurement in association with uterine artery Doppler as a screening too for placental insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hypertension under medication
* Diabetes
* Thrombophilia
* Previous history of pre-eclampsia
* Previous history of unexplained stillbirth
* Previous history of placental abruption
* Previous history of SGA (< 10th centile)
* History of pre-eclampsia or chronic hypertension before 45 years in the mother or a sister
* Obesity (BMI>30)
* Nulliparous after 40 years
* Assisted conception with donor

Exclusion Criteria:

* Multiple pregnancy
* Complicated pregnancy with a high probability of required fetal extraction before term
* Pregnancy requiring termination
* Unability to understand the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women at increased risk of pre-eclampsia (PE) and intrauterine growth restriction (IUGR)
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2003-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franck Perrotin, MD-PhD, Principal Investigator — Tours University Hospital
Locations (1):
- Olympe de Gouges Women Health Centre, Bretonneau University Hospital, Tours, France

REFERENCES:
- [Background] Papageorghiou AT, Leslie K. Uterine artery Doppler in the prediction of adverse pregnancy outcome. Curr Opin Obstet Gynecol. 2007 Apr;19(2):103-9. doi: 10.1097/GCO.0b013e32809bd964. PMID 17353676
- [Background] Guven MA, Ertas IE, Kilinc M, Coskun A, Ekerbicer H. Combining mid-trimester maternal plasma homocysteine with uterine artery doppler velocimetry: is it useful? Arch Gynecol Obstet. 2007 Jun;275(6):439-43. doi: 10.1007/s00404-006-0281-5. Epub 2006 Nov 17. PMID 17111155
- [Background] Spencer K, Yu CK, Savvidou M, Papageorghiou AT, Nicolaides KH. Prediction of pre-eclampsia by uterine artery Doppler ultrasonography and maternal serum pregnancy-associated plasma protein-A, free beta-human chorionic gonadotropin, activin A and inhibin A at 22 + 0 to 24 + 6 weeks' gestation. Ultrasound Obstet Gynecol. 2006 Jun;27(6):658-63. doi: 10.1002/uog.2676. PMID 16493628
- [Background] Tommaselli GA, Pighetti M, Nasti A, D'Elia A, Guida M, Di Carlo C, Bifulco G, Nappi C. Serum leptin levels and uterine Doppler flow velocimetry at 20 weeks' gestation as markers for the development of pre-eclampsia. Gynecol Endocrinol. 2004 Sep;19(3):160-5. doi: 10.1080/09513590400007267. PMID 15697078